CLINICAL TRIAL: NCT00003939
Title: Phase II Study on ET-743 in Advanced Soft Tissue Sarcomas of the Adult
Brief Title: Ecteinascidin 743 in Treating Patients With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-62982-16993; EORTC-62982
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors; Endometrial Cancer; Gastrointestinal Stromal Tumor; Ovarian Cancer; Sarcoma; Small Intestine Cancer
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; small intestine leiomyosarcoma; adult alveolar soft-part sarcoma; adult epithelioid sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult rhabdomyosarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; uterine carcinosarcoma; uterine leiomyosarcoma; endometrial stromal sarcoma; ovarian sarcoma; adult meningeal hemangiopericytoma; gastrointestinal stromal tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Endometrial Neoplasms; Gastrointestinal Stromal Tumors; Ovarian Neoplasms; Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Sarcoma, Alveolar Soft Part; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Rhabdomyosarcoma; Sarcoma, Endometrial Stromal | interventions — Trabectedin

INTERVENTIONS:
Drug: trabectedin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ecteinascidin 743 in treating patients who have advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the therapeutic activity of ecteinascidin 743 in patients with advanced soft tissue sarcomas. II. Determine the duration of response in these patients. III. Determine the acute side effects in these patients.

OUTLINE: This is a multicenter study. Patients receive ecteinascidin 743 (ET-743) IV over 24 hours every 3 weeks. Treatment continues for at least 2-6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks until disease progression and every 12 weeks after disease progression.

PROJECTED ACCRUAL: Approximately 28-44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven soft tissue sarcoma, including the following cell types: Malignant fibrous histiocytoma Liposarcoma Rhabdomyosarcoma Synovial sarcoma Malignant paraganglioma Fibrosarcoma Leiomyosarcoma Angiosarcoma including hemangiopericytoma Neurogenic sarcoma Unclassified sarcoma Miscellaneous sarcoma including mixed mesodermal tumors of the uterus Cell types NOT allowed: Malignant mesothelioma Chondrosarcoma Neuroblastoma Osteosarcoma Ewing's sarcoma Embryonal rhabdomyosarcoma Measurable lesion with evidence of progression within 6 weeks prior to study (osseous lesions, hepatomegaly, lymphedema, ascites, and pleural lesions are not considered measurable) No symptomatic or known CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: Neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.75 mg/dL Albumin at least 2.5 g/dL AST and ALT less than 1.5 times upper limit of normal (ULN) (2.5 times ULN if liver metastasis present) Alkaline phosphatase less than 2.5 times ULN No other significant hepatic disease (e.g., active hepatitis, cirrhosis, etc.) Renal: Creatinine no greater than 1.36 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No prior cardiovascular disease Other: No other severe medical illness No psychosis No prior or concurrent second primary malignant tumors, except adequately treated carcinoma in situ of the cervix or basal cell carcinoma Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy No more than 1 prior regimen of combination chemotherapy OR No more than 2 prior single agent regimens No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to sole index lesion No concurrent radiotherapy Surgery: Not specified Other: No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Primary Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Le Cesne, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris

REFERENCES:
- [Background] Therasse P, Le Cesne A, Van Glabbeke M, Verweij J, Judson I; EORTC Soft Tissue and Bone Sarcoma Group. RECIST vs. WHO: prospective comparison of response criteria in an EORTC phase II clinical trial investigating ET-743 in advanced soft tissue sarcoma. Eur J Cancer. 2005 Jul;41(10):1426-30. doi: 10.1016/j.ejca.2005.04.005. PMID 15919202
- [Result] Le Cesne A, Blay JY, Judson I, Van Oosterom A, Verweij J, Radford J, Lorigan P, Rodenhuis S, Ray-Coquard I, Bonvalot S, Collin F, Jimeno J, Di Paola E, Van Glabbeke M, Nielsen OS. Phase II study of ET-743 in advanced soft tissue sarcomas: a European Organisation for the Research and Treatment of Cancer (EORTC) soft tissue and bone sarcoma group trial. J Clin Oncol. 2005 Jan 20;23(3):576-84. doi: 10.1200/JCO.2005.01.180. PMID 15659504
- [Result] Blay JY, Le Cesne A, Verweij J, Scurr M, Seynaeve C, Bonvalot S, Hogendoorn P, Jimeno J, Evrard V, van Glabbeke M, Judson I. A phase II study of ET-743/trabectedin ('Yondelis') for patients with advanced gastrointestinal stromal tumours. Eur J Cancer. 2004 Jun;40(9):1327-31. doi: 10.1016/j.ejca.2004.02.005. PMID 15177491
- [Result] Le Cesne A, Judson I, Blay JY, et al.: Phase II study of ET-743 in advanced soft tissue sarcoma (ASTS) in adults: a STBSG-EORTC trial. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A-2182, 2000.